CLINICAL TRIAL: NCT04024969
Title: DECISIve - DiagnosE Using the Central veIn SIgn. A Prospective Diagnostic Superiority Study Comparing T2* MRI and Lumbar Puncture in Patients Presenting With Possible Multiple Sclerosis
Brief Title: DiagnosE Using the Central veIn SIgn
Acronym: DECISIve
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18GNS004
Record Dates: First submitted 2019-06-12; First posted 2019-07-18 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2019-07

CONDITIONS: Multiple Sclerosis
Keywords: Central Vein Sign; Translational Neuroimaging; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Magnetic Resonance Myelography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinically isolated syndrome: Those presenting for diagnositic evaluation of multiple sclerosis, not currently meeting the 2017 McDonald criteria.
  Interventions: Diagnostic Test: T2* MRI; Diagnostic Test: Lumbar puncture to test for presence of unmatched oligoclonal bands

INTERVENTIONS:
Diagnostic Test: T2* MRI — Research T2* weighted MRI sequence
Diagnostic Test: Lumbar puncture to test for presence of unmatched oligoclonal bands — Current clinical standard practice

SUMMARY:
There is currently no agreement on the best way to diagnose Multiple Sclerosis (MS). Frequently, people suspected of having MS have a standard MRI scan and undergo a 'lumbar puncture' (a thin needle is inserted between the bones in the lower spine). Patients often report they find it painful and it can cause unintended complications requiring hospitalisations or time off work to recover.

Although the fluid taken during a lumbar puncture can show evidence of disease, this is not always the case. Doctors do not find abnormalities in everyone who has MS but some people with conditions that can mimic MS, but need very different treatment, have similar lumbar puncture abnormalities. Both of these problems can lead to misdiagnosis.

A new MRI scan allows doctors to see small veins that run through damaged areas of the brain in people with MS. It has been shown that this is a specific finding to MS, seldom seen in other conditions. It is not painful and carries few or no risks.

This research aims to change the way people are diagnosed with MS and reduce the number of lumbar punctures used. The investigators will recruit a large number of people from different hospitals whose doctors suspect they may have MS. They will be invited to have the new eight-minute MRI scan. After 18 months, the investigators will find out what diagnosis is eventually reached and compare this to the finding of the new scan. The investigators will then compare the accuracy, speed, costs and acceptability of the different tests needed to make a diagnosis of MS and establish if most lumbar punctures can be replaced by a slightly longer MRI scan. This research could provide the National Health Service with a scientific approach to diagnose MS which is safer, more cost effective and importantly, more acceptable to patients.

DETAILED DESCRIPTION:
The North American Imaging in MS Cooperative has reviewed the utility of the central vein sign (CVS) in the diagnosis of MS in 2015. They concluded that "To formally establish the clinical value of the CVS for the differential diagnosis at disease onset, a large, prospective, multicentre study including patients at first presentation of possible MS is necessary". The paper outlining the 2017 McDonald diagnostic criteria for MS specifically mentions the promise of the CVS but suggests that it "requires detailed investigation to determine whether it is useful and practical". The rationale of this study is to provide an overwhelming case for a straightforward and rapid clinical adoption of our MRI test, which will change our ability to confirm or refute the diagnosis of MS.

Radiologists and neurologists can also readily interpret our proposed CVS using a simple 'rule of six' that was described in a previous study. This involves the detection of any six lesions with a central vein present. This rule has the potential to be easily implemented in clinical practice if it has superior diagnostic sensitivity, when compared to lumbar puncture results.

If the CVS can be shown to have superior diagnostic sensitivity at first presentation of MS, when compared to performing a lumbar puncture, then lumbar punctures can be avoided in many patients. These patients will benefit in several ways. The patients will avoid a procedure that is often painful or unpleasant. Those who currently refuse to have lumbar puncture will benefit from expedited diagnosis, limiting their anxiety and uncertainty. A secure diagnosis could lead to more rapid treatment decisions and a better long-term prognosis. In addition, fewer workdays will be lost attending hospital for investigation. From the NHS' perspective, it would avoid day case hospital admissions for lumbar punctures and readmissions to treat the common complication of post lumbar puncture headaches. This would create significant cost savings, when considering the significant number of patients undergoing this diagnostic process.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years.
2. Presentation with a typical clinically isolated syndrome (Thompson et al. 2017) for diagnostic evaluation of MS.

Exclusion Criteria:

1. Fulfils the diagnosis of MS, as defined by the 2017 revision of McDonald diagnostic criteria (Thompson et al. 2017).
2. Unwilling or unable to comply with the requirements of this protocol including the presence of any condition (physical, mental, or social) that, in the opinion of the PI, is likely to affect the participant's ability to comply with the study protocol.
3. Unable to provide informed consent.
4. Contraindication or inability to undergo MRI due to metal or metal implants, pregnancy, claustrophobia, pain, spasticity, or excessive movement related to tremor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Most participants are expected to have been evaluated by a hospital doctor (usually neurologist or ophthalmologist) at the local site and referred for diagnostic testing to the local MS team.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2019-11-06 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of the central vein sign (CVS) on T2* MRI scan and lumbar puncture with oligoclonal band testing at diagnosing MS at the time of the patients' first presentation. | 18 months
  The reference standard for both tests will be clinical diagnosis 18 months after recruitment. The sensitivity of each test will be reported separately along with 95% confidence intervals. The sensitivity of the tests will be compared using McNemar's test for paired proportions.

SECONDARY OUTCOMES:
The specificity of the central vein sign (CVS) on T2* MRI scan and lumbar puncture with oligoclonal band testing at diagnosing MS at the time of the patients' first presentation. | 18 months
  The reference standard for both tests will be clinical diagnosis 18 months after recruitment. The specificity of each test will be reported separately along with 95% confidence intervals. The specificity of the tests will be compared using McNemar's test for paired proportions.
The sensitivity and specificity of the 'rule of six' proposed in Mistry et al. 2016. | 18 months
  The reference standard for the test will be clinical diagnosis 18 months after recruitment. The sensitivity and specificity of the 'rule of six' test will be reported separately along with 95% confidence intervals. The sensitivity and specificity of the 'rule of six' against lumbar puncture result will be compared using McNemar's test for paired proportions.

OTHER OUTCOMES:
The percentage agreement between blinded raters of the CVS amongst different observers. | 18 months
  The receiver operating characteristic curve for T2* MRI will be presented along with percentage agreement between blinded raters.
The sensitivity and specificity of combing the CVS with the results of the lumbar puncture. | 18 months
  The reference standard for the test will be clinical diagnosis 18 months after recruitment. The sensitivity and specificity of a positive result in either the CVS or lumbar puncture result will be reported separately along with 95% confidence intervals.
A sensitivity analysis, allowing for variation in test performance between sites, using a mixed effects logistic regression model. | 18 months
  A review of whether there is evidence of test performance variability when performed at different hospitals.
The sensitivity and specificity of the 3D FLAIR* (a research imaging technique) | 18 months
  The reference standard for the test will be clinical diagnosis 18 months after recruitment. The sensitivity and specificity of 3D FLAIR* will be reported separately along with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Evangelou, MD, Principal Investigator — Clinical Neurology, Division of Clinical Neuroscience, University of Nottingham
Locations (4):
- United Kingdom (4):
  - Cardiff & Vale University Lhb, Cardiff
  - Barts Health Nhs Trust, London
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals Nhs Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Mistry N, Abdel-Fahim R, Samaraweera A, Mougin O, Tallantyre E, Tench C, Jaspan T, Morris P, Morgan PS, Evangelou N. Imaging central veins in brain lesions with 3-T T2*-weighted magnetic resonance imaging differentiates multiple sclerosis from microangiopathic brain lesions. Mult Scler. 2016 Sep;22(10):1289-96. doi: 10.1177/1352458515616700. Epub 2015 Dec 10. PMID 26658816